CLINICAL TRIAL: NCT02518724
Title: The Effect of Remote Ischemic Preconditioning (RIPC) on Physical Performance and Exertional Rhabdomyolysis
Brief Title: The Effect of Remote Ischemic Preconditioning on Physical Performance and Exertional Rhabdomyolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SHEBA-15-2139-OF-CTIL
Record Dates: First submitted 2015-07-13; First posted 2015-08-10 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Physical Performance; Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC intervention group (Active Comparator): The experiment protocol consist 2 series (with a month between them), both series include the described 3 days:
  Day 1 - anthropometry measurements and VO2max test (BRUCE protocol). Day 2 - steps test (heled protocol). Day 3 - anaerobic test (wingate protocol), 1 hour rest and time to exhaustion test (heled protocol).
  the second series will be performed after RIPC intervention exposure at the beginning of every meeting.
  Interventions: Procedure: RIPC intervention exposure
- false exopsure group (Placebo Comparator): The experiment protocol consist 2 series (with a month between them), both series include the described 3 days:
  Day 1 - anthropometry measurements and VO2max test (BRUCE protocol). Day 2 - steps test (heled protocol). Day 3 - anaerobic test (wingate protocol), 1 hour rest and time to exhaustion test (heled protocol).
  the second series will be performed after placebo intervention exposure at the beginning of every meeting.
  Interventions: Procedure: placebo intervention exposure

INTERVENTIONS:
Procedure: RIPC intervention exposure — placing a sphygmomanometer on the non-dominant hand and applying pressure of 200 mmHg for 5 min followed by 5 min without pressure X 4 repeats
  Arms: RIPC intervention group
Procedure: placebo intervention exposure — placing a sphygmomanometer on the non-dominant hand and applying pressure of 100 mmHg for 5 min followed by 5 min without pressure X 4 repeats.
  Arms: false exopsure group

SUMMARY:
In order to examine the effect of RIPC on skeleton muscle exertional damage and on aerobic and anaerobic physical performances, 30 healthy volunteers will undergo a series of different physical tests twice; once without intervention and a second time with RIPC intervention or placebo (false) intervention.

DETAILED DESCRIPTION:
30 healthy civilians volunteers will be recruited and divided randomly into 2 groups: RIPC group and control group.

The experiment protocol consist 2 series (with a month between them), both series include the described 3 days:

Day 1 - anthropometry measurements and VO2max test (BRUCE protocol). Day 2 - steps test (heled protocol). Day 3 - anaerobic test (wingate protocol), 1 hour rest and time to exhaustion test (heled protocol).

The first series will be performed without applying any intervention and is considered as baseline measurements for both groups. the second series will be performed as follows: a. RIPC group: applying RIPC exposure (placing a sphygmomanometer on the non-dominant hand and applying pressure of 200 mmHg for 5 min followed by 5 min without pressure X 4 repeats) at the beginning of every meeting. b. control group: with placebo (false) exposure (placing a sphygmomanometer on the non-dominant hand and applying pressure of 100 mmHg for 5 min followed by 5 min without pressure X 4 repeats) at the beginning of every meeting.

Blood ample, lactic acid and urine sample will be tested at the beginning and end of every meeting (testing for muscle, skeleton and kidney function markers).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30
* healthy civilians volunteers
* with no background illnesses
* above average fitness

Exclusion Criteria:

* known chronic medical illness
* routine medication usage
* history of rhabdomyolysis
* the physician decision

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
creatine phosphokinase (CPK) | 6 experiment days for each participant
  CPK is a marker for muscle damage assessed in blood test. blood sample will be taken before and after step test, anaerobic test and time to exhaustion test.

SECONDARY OUTCOMES:
oxygen consumption (VO2) | 6 experiment days for each participant
  VO2 will be monitored continuously using a metabolic system (ERGOTEST 680, ZAN, GERMANY ) during VO2max test and time to exhaustion test
heart rate variability (HRV) | 6 experiment days for each participant
  HRV will be measured using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch) at rest for 10 min, before and after RIPC. data will be analysed by an expert.
lactic acid | 6 experiment days for each participant
  lactic acid level is assessed from blood drop (finger sting), will be taken before and after every test. lactic acid is a marker for anaerobic effort evaluating.
blood count | 6 experiment days for each participant
  blood counts are done to monitor overall health and to confirm a diagnosis of some medical conditions.
apolipoprotein A1 (APO-A1) levels | 6 experiment days for each participant
  APO-A1 is measured in blood chemistry as a marker for cholesterol.
renal function (composite) | 6 experiment days for each participant
  renal function (in order or not) will be evaluated from two markers measured in blood sample (chemistry): creatinine and urea.
inflammation (composite) | 6 experiment days for each participant
  C-reactive protein (CRP) and blood sedimentation rate (assessed from blood sample) are indicators for inflammation.
heart rate | 6 experiment days for each participant
  HR will be monitored during the physical tests using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel